CLINICAL TRIAL: NCT04741165
Title: An Open-label, Multicenter, Phase II Clinical Study of HX008 in Combination With Bevacizumab or Lenvatinib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Brief Title: Study of HX008 in Combination With Bevacizumab or Lenvatinib for the Treatment of Advanced Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX008-II-HCC-01
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: HX008+Bevacizumab (Experimental): Participants receive HX008 200 mg intravenous (IV) every 3 weeks (Q3W) plus bevacizumab 15 mg/kg, IV, Q3W.
  Interventions: Drug: HX008; Drug: Bevacizumab
- Experimental: HX008+Lenvatinib (Experimental): Participants receive HX008 200 mg intravenous (IV) every 3 weeks (Q3W) plus lenvatinib 12 mg (for participants with screening body weight ≥60 kg) or 8 mg (for participants with screening body weight <60 kg) orally once a day (QD).
  Interventions: Drug: HX008; Drug: Lenvatinib

INTERVENTIONS:
Drug: HX008 — 200 mg administered as IV infusion on Day 1 of each 21-day cycle.
Drug: Bevacizumab — 15 mg/kg administered as IV infusion on Day 1 of each 21-day cycle.
  Other Names: AVASTIN®
  Arms: Experimental: HX008+Bevacizumab
Drug: Lenvatinib — Administered orally once a day during each 21-day cycle
  Other Names: LENVIMA®
  Arms: Experimental: HX008+Lenvatinib

SUMMARY:
This is a multi-center,open-label study to evaluate the efficacy and safety of anti-PD-1 antibody HX008 plus bevacizumab or lenvatinib in the first-line treatment of patients with unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Understood and signed an informed consent form.
* Age ≥ 18 and ≤ 75 years old, male or female.
* Has histologically- or cytologically-confirmed diagnosis of unresectable hepatocellular carcinoma.
* Has Barcelona Clinic Liver Cancer (BCLC) Stage C disease, or BCLC Stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach.
* Child-Pugh class A and B (≤7 points).
* Has not received any systematic treatment for HCC.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Score.
* Life expectancy ≥ 3 months.
* Has at least one measurable disease based on RECIST 1.1.
* Has adequate organ function as defined in the protocol.
* Female participants of childbearing potential should have a negative pregnancy within 7 days before the randomization. Male and female participants should agree to use an adequate method of contraception during the experiment and 1 year after the last administration of the test drugs.

Exclusion Criteria:

* Histologically or cytologically documented fibrolamellar hepatocellular carcinoma, sarcoma-like hepatocellular carcinoma, cholangiocarcinoma, etc.
* Diagnosed additional malignancy within 3 years prior to the first dose of trial, with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin,curatively resected in situ cervical or non-muscle invasive bladder cancers.
* Has received locoregional therapy or surgery within 4 weeks prior to the first dose of trial treatment; received palliative radiotherapy or herbal medicine within 2 weeks prior to the first dose of trial treatment;
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* HBV-DNA>2000 IU/mL or 10^4 copy/mL; HCV-RNA>10^3 copy/mL.
* Has had esophageal or gastric variceal bleeding within the last 6 months.
* Portal vein tumor thrombus (PVTT) involves both the main trunk and contralateral branch or upper mesenteric vein. Inferior vena cava tumor thrombus.
* Other obvious hemorrhagic tendency or evidence on important coagulation disorder.
* Serious cardiovascular and cerebrovascular diseases.
* Inability to swallow tablets, malabsorption syndrome or any other condition that affects gastrointestinal absorption.
* Serious, uncured wound, active ulcer or untreated bone fracture.
* Uncontrolled pericardial effusion, uncontrolled pleural effusion or clinically obvious moderate peritoneal effusion at screening.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Has received a major surgery within 4 weeks prior to the first dose of tiral treatment.
* Has received system treatment with corticosteroids (dose >10mg/day prednison or other therapeutic hormones) within 2 weeks prior to the first dose of trial treatment.
* Has a history of non-infectious pneumonitis that required steroids or has current pneumonitis.
* Has known active tuberculosis (Bacillus tuberculosis)
* Has a history of testing positive for human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS), or stem cell transplantation or organ transplantation.
* Co-infection of HBV and HCV.
* Any serious acute and chronic infection within 4 weeks prior to the first dose of trial treatment, or infection requiring systemic antibacterial, antifungal or antiviral therapy within 2 weeks prior to the first dose of trial treatment.
* Has participated in other anticancer drug clinical trials within 4 weeks.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 15 months
  ORR was defined as the percentage of participants who have a complete response (CR) or a partial response (PR), per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to approximately 15 months
  DCR was defined as the percentage of participants who have a CR or a PR or a stable disease (SD), per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.
Duration of Response (DOR) | up to approximately 15 months
  DOR was defined as the time from the first documented evidence of a response of CR or PR, per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by investigators.
Progression-free Survival (PFS) | up to approximately 15 months
  PFS was defined as the time from randomization to the first documented disease progression per RECIST 1.1 assessed by investigators or death due to any cause, whichever occurs first.
Overall Survival (OS) | up to approximately 20 months
  OS was defined as the time from the date of beginning of HX008 administration until date of death from any cause.
Time to Disease Progression (TTP) | up to approximately 15 months
  TTP is defined as the time from randomization to the first documented disease progression per RECIST 1.1 as assessed by investigators.
Number of participants with adverse events (AEs) | up to approximately 20 months
  An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product temporally associated with the use of study treatment, whether or not considered related to the study treatment

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - The Fist Affiliated Hospital of USTC(Anhui Provincial hospital), Hefei, Anhui
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Yuhe Integrated Traditional Chinese and Western Medicine Rehabilitation Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, shenzhen center, Shenzhen, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The First Affiliated University of Nanhua University, Hengyang, Hunan
  - The Sixth People's Hospital of Shenyang, Shenyang, Liaoning
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality
  - The Central Hospital of Lishui City, Lishui, Zhejiang